CLINICAL TRIAL: NCT00732095
Title: Promoting Self-Change From Alcohol Problems: Mechanisms of Change in a Community-Based Intervention
Acronym: PSC3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nova Southeastern University (Other)
Responsible Party: Nova SEU University, Dr. Linda C.S
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R21AA017136 (NIH); 1R21AA017136 (NIH)
Record Dates: First submitted 2008-08-07; First posted 2008-08-11 (Estimated); Last update posted 2010-12-14 (Estimated); Status verified 2010-12

CONDITIONS: Alcohol Drinking; Alcohol Abuse
Keywords: Self-change; Natural recovery; Alcohol Drinking; Mechanisms of Change; Advertisements
MeSH Terms: conditions — Alcohol Drinking; Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental (Experimental): Immediate Ad
  Interventions: Behavioral: Promoting Self-Change with Ads

INTERVENTIONS:
Behavioral: Promoting Self-Change with Ads — Use of Ads immediate or delayed or no ad

SUMMARY:
Research has found that natural recovery (self-change) is a very common pathway to change for individuals with alcohol problems, accounting for nearly 75% of recoveries in several national surveys.

Although few members of the public are aware that self-change is possible, it also is the case that many individuals with alcohol problems do not enter treatment because of the stigma or fear of being labeled. The proposed study is based on findings from a recent randomized controlled trial designed to promote self-change in the community for problem drinkers who had never been in treatment. Media advertisements were used to recruit 825 participants. Eligible respondents were sent assessment materials to complete. After the assessment materials were returned, participants were randomly assigned to receive two alcohol pamphlets that were freely available in the community or personalized feedback based on their assessment responses (e.g., how their drinking compared to national norms, health risks associated with their drinking). A 1-year follow up found that while there were no differences in drinking behavior between the groups, both groups had very substantial reductions in their drinking 1-year pre- to 1-year post-intervention. In an attempt to determine what accounted for the change, participants' reports of their drinking were evaluated with regard to critical study elements (e. g., when assessment materials were received). Surprisingly, results revealed that many changed after seeing the advertisement, and before receiving the assessment materials to complete. This suggests that either seeing the ad ("Thinking about changing your drinking?") or a message in the ad ("Did you know that 75% of people change their drinking on their own?") may have catalyzed the change. To evaluate when change occurs and the mechanisms that may give rise to change, a randomized controlled trial involving 3 groups will be conducted. The groups will differ in whether they receive a message informing them that self-change is a common phenomenon (two groups will receive the message, one will not) and the occasion when the message is delivered (consenting to the study and before the assessment vs. with the intervention material). Comparisons made possible by the experimental design will allow an evaluation of the message as a precipitant of change. The use of Timeline Followback retrospective reports of daily drinking and recording of critical dates will allow statistical analysis of patterns of inflection (i.e., change in drinking) related to seeing the ad, receiving the message, receiving and completing the assessment materials, and receiving the intervention materials. Possible explanations for how the message could function as a mechanism of behavior change are offered (e.g., catastrophe theory, cognitive social learning theory). The ultimate objective of this research is to develop cost-effective, large scale interventions that can be viewed as an early stage in a public health, stepped care model by encouraging self-change for individuals with alcohol problems.

DETAILED DESCRIPTION:
Brief Overview: Research has found that natural recovery (self-change) is a very common pathway to change for individuals with alcohol problems, accounting for nearly 75% of recoveries in several national surveys. Although few members of the public are aware that self-change is possible, it also is the case that many individuals with alcohol problems do not enter treatment because of the stigma or fear of being labeled. The proposed study is based on findings from a recent randomized controlled trial designed to promote self-change in the community for problem drinkers who had never been in treatment. Media advertisements were used to recruit 825 participants. Eligible respondents were sent assessment materials to complete. After the assessment materials were returned, participants were randomly assigned to receive two alcohol pamphlets that were freely available in the community or personalized feedback based on their assessment responses (e.g., how their drinking compared to national norms, health risks associated with their drinking). A 1-year follow up found that while there were no differences in drinking behavior between the groups, both groups had very substantial reductions in their drinking 1-year pre- to 1-year post-intervention. In an attempt to determine what accounted for the change, participants' reports of their drinking were evaluated with regard to critical study time points (e. g., when assessment materials were received). Surprisingly, results revealed that many changed after seeing the advertisement, and before receiving the assessment materials to complete. This suggests that either seeing the ad ("Thinking about changing your drinking?") or a message in the ad ("Did you know that 75% of people change their drinking on their own?") may have catalyzed the change. To evaluate when change occurs and the mechanisms that may give rise to change, a randomized controlled trial involving 3 groups will be conducted. The groups will differ in whether they receive a message informing them that self-change is a common phenomenon (two groups will receive the message, one will not) and the occasion when the message is delivered (consenting to the study and before the assessment vs. with the intervention material). Comparisons made possible by the experimental design will allow an evaluation of the message as a precipitant of change. The use of Timeline Followback retrospective reports of daily drinking and recording of critical dates will allow statistical analysis of patterns of inflection (i.e., change in drinking) related to seeing the ad, receiving the message, receiving and completing the assessment materials, and receiving the intervention materials. Possible explanations for how the message could function as a mechanism of behavior change are offered (e.g., catastrophe theory, cognitive social learning theory). The ultimate objective of this research is to develop cost-effective, large scale interventions that can be viewed as an early stage in a public health, stepped care model by encouraging self-change for individuals with alcohol problems.

Main Goals and Justification The proposed research project is an outgrowth and extension of research Drs. Linda and Mark Sobell have been conducting for many years. That research began with investigations of individuals who recovered from alcohol problems without treatment (natural recoveries). A major finding of the natural recovery research, conducted in Canada but now supported by similar data from the US, was that rather than an uncommon occurrence, self-change is the major pathway to change. Another finding of our natural recovery research was that the most commonly reported precipitant of change was a cognitive appraisal (i.e., cost-benefit analysis) 1that occurred over time rather than some particular isolated event (event-precipitated recovery). The individuals most likely to achieve a natural recovery are those who do not have severe problems and who also tend not to access treatment resources.

Our natural recovery research findings led to the design of a study, Promoting Self-Change, intended to encourage problem drinkers within a community setting who have never sought treatment or formal help to change their drinking their own (Sobell et al., 1996). The experimental intervention in the PSC study was modeled on the evidence-based materials developed for use in the Guided Self-Change model of treatment, a brief cognitive-behavioral motivational intervention Although both the experimental and control groups showed significant reduction in their drinking from 1-year pre- to 1-year post-intervention, the results showed that people who received the experimental motivational materials showed no greater change than those who received the two alcohol pamphlets that were freely available in the community (Sobell et al., 2002).

Fortunately, because we had collected drinking data using the Timeline Followback (Sobell & Sobell, 1992, 2003, 2007 in press) and kept records of important events (e.g., date person called to be screened, date assessment materials mailed), it allowed us to explore when change occurred. Contrary to the our hypothesis, the major reduction in drinking does not appear to have occurred after the intervention materials were received, but rather after participants saw the study advertisements. Thus, as will be discussed in detail in the design section, seeing the ads and the message in the ads was identified as possible important precipitants of change. The proposed project is a randomized controlled study to investigate these issues.

Based on our previous Promoting Self-Change study, we will conduct a randomized controlled trial consisting of three groups and designed to tease apart alternative possible explanations of mechanisms of behavior change within a community based mail intervention. In particular, the study will investigate the timing of points of inflection (i.e., change) in participants' reported drinking as they participate in the study. The three experimental groups will differ in whether they receive a message informing them that self-change is a common phenomenon (two groups will receive the message, one will not) and the occasion when the message is delivered (when consenting to the study and before the assessment vs. with the intervention material). This design allows the following 5 objectives to be addressed:

* To evaluate if a message that communicates that self-change (i.e., alcohol problem) is common will prompt participants to engage in a process of self-change resulting in changes in their drinking behavior
* To evaluate whether there is a difference in effectiveness depending on when the message that self-change is common is presented (before the assessment versus at the intervention)
* To evaluate whether only seeing an advertisement prompts participants to think about changing their drinking and then change on their own in the absences of a message that self-change is common
* To evaluate whether receiving the message as part of the intervention materials adds value over the effect of receiving only the intervention materials.
* To conduct correlative investigations of whether participants report changes in their drinking contiguous with first seeing the advertisement, receiving the assessment materials (without the message), and receiving the intervention feedback.

Possible explanations for how the message could function as a mechanism of behavior change are offered from catastrophe theory and cognitive social learning theory. The ultimate objective of this line of research is the development of cost-effective, large scale interventions that can serve as an early stage in a public health, stepped care model by encouraging self-change in the community for individuals with alcohol problems.

ELIGIBILITY:
Inclusion Criteria:

* 21 years of age or older (legal drinking age in US)
* report drinking an average of >12 drinks per week or having consumed ≥ 5 drinks on ≥ 5 days in the past year
* sign an informed consent
* willing to participate in a 90-day follow-up interview by mail after the intervention
* willing to provide the name, address and phone number of a relative or friend who has known the participant and is willing to be provide information in the form of a short questionnaire about the participant's alcohol use and functioning 90 days after the intervention starts

Exclusion Criteria:

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 283 (Actual)
Dates: Start 2008-03; Primary Completion 2010-05 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
reduced alcohol use | 3 months post intervention

SECONDARY OUTCOMES:
reduced alcohol related consequences | 3 months post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Linda C Sobell, Ph.D., Principal Investigator — Nova Southeastern University
Locations (1):
- Nova Southeastern University, Center for Psychological Studies, Fort Lauderdale, Florida, United States

REFERENCES:
- [Background] Sobell LC, Sobell MB, Leo GI, Agrawal S, Johnson-Young L, Cunningham JA. Promoting self-change with alcohol abusers: a community-level mail intervention based on natural recovery studies. Alcohol Clin Exp Res. 2002 Jun;26(6):936-48. PMID 12068264